CLINICAL TRIAL: NCT01821365
Title: End Tidal Carbon Dioxide Monitoring for Evaluating Changes of Arterial Carbon Dioxide After Noninvasive Mechanical Ventilation in Chronic Obstructive Pulmonary Disease
Brief Title: End Tidal Carbon Dioxide Monitoring for Evaluating Changes of PaCO2 After Noninvasive Mechanical Ventilation in COPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, ting Jiang, MM, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: 2009CB522100
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: COPD
Keywords: COPD,PETCO2,PaCO2
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Sidestream end-tidal CO2 has been found to be closely correlated to PaCO2 especially when people have the stable hemodynamics and normal lung function. PETCO2 can basically reflect the level of PaCO2,but some investigators found that PETCO2 measurements did not reflect PaCO2 in COPD patients.There may be several reasons for this discrepancy. Due to airway obstruction and ventilation-perfusion mismatch, there is a delay in the maximum alveolar concentration of CO2 reaching the cannula, which may give lower PETCO2 values compared with PaCO2. To overcome this disadvantage, we tried to prolong their expiratory time (extend to 5-8s) in order to guarantee adequate time for alveolar CO2 reaching the cannula.our study mainly focus on two issues.First, to explore the optimal depth of tube placed when patients with COPD breathe spontaneously or receive noninvasive ventilation, and compare the differences of two condition at the same time. Secondly, to evaluate the agreement between the PaCO2 and sidestream PETCO2（5s）values in COPD patients receiving noninvasive ventilation when our extension tube locates in the optimal position, and investigate whether PETCO2（5s）can be used to monitor ventilation status dynamically.

DETAILED DESCRIPTION:
Non-invasive positive pressure ventilation(NPPV) can significantly improve gas exchange and relieve respiratory muscle fatigue for COPD,and arterial blood gas is the gold standard to evaluate ventilation status,but the procedure is time consuming,invasive, painful and in some patients.

Sidestream end-tidal CO2 has been found to be closely correlated to PaCO2 especially when people have the stable hemodynamics and normal lung function. PETCO2 can basically reflect the level of PaCO2, but for patients with COPD, due to the presence of airway obstruction and emphysema formation, which cause ventilation-perfusion ratio(V/Q) , result to dead space-tidal volume ratio(VD/VT) and right-to-left shunting(Qs/Qt), the time of various lung units discharge of carbon dioxide is not synchronous. Some investigators found that PETCO2 measurements did not reflect PaCO2 in COPD patients. There may be several reasons for this discrepancy. Due to airway obstruction and ventilation-perfusion mismatch, there is a delay in the maximum alveolar concentration of CO2 reaching the cannula, which may give lower PETCO2 values compared with PaCO2. To overcome this disadvantage, we tried to prolong their expiratory time (extend to 5-8s) in order to guarantee adequate time for alveolar CO2 reaching the cannula.

our study mainly focus on two issues.First, to explore the optimal depth of tube placed when patients with COPD breathe spontaneously or receive noninvasive ventilation, and compare the differences of two condition at the same time. Secondly, to evaluate the agreement between the PaCO2 and sidestream PETCO2（5s）values in COPD patients receiving noninvasive ventilation when our extension tube locates in the optimal position, and investigate whether PETCO2（5s）can be used to monitor ventilation status dynamically.

ELIGIBILITY:
Inclusion Criteria:1.patients are enrolled in accordance with 2011 international treatment guidelines of COPD.

2.patients are in a clear state of mind and can incompliance with clinicians to extend breathing only using nose and closing mouth.

Exclusion Criteria:1.Hemodynamic instability. 2.Pulmonary embolism,Pneumothorax, pleural effusion, upper airway obstruction,Chest trauma, chest wall deformities, neuromuscular diseases, lung tumor.

3.combinating acute exacerbation of bronchial asthma in this hospitalization. 4.Nose and mouth trauma, deformity, or recent surgery.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a COPD exacerbation who admitted to the respiratory department of First Affiliated Hospital of Guangzhou Medical University,Guangzhou,Guangdong,China
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
the agreement and correlation between the partial pressure of end-tidal carbon dioxide(PETCO2) | one day
  PETCO2 was measured by using sidestream capnometer though prolonged expiratory method(extend to 5s) , and obtained arterial blood sampling simultaneously.

CONTACTS AND LOCATIONS:
Overall Officials: Rongchang Chen, MD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Wu CH, Chou HC, Hsieh WS, Chen WK, Huang PY, Tsao PN. Good estimation of arterial carbon dioxide by end-tidal carbon dioxide monitoring in the neonatal intensive care unit. Pediatr Pulmonol. 2003 Apr;35(4):292-5. doi: 10.1002/ppul.10260. PMID 12629627
- [Result] Trevisanuto D, Giuliotto S, Cavallin F, Doglioni N, Toniazzo S, Zanardo V. End-tidal carbon dioxide monitoring in very low birth weight infants: correlation and agreement with arterial carbon dioxide. Pediatr Pulmonol. 2012 Apr;47(4):367-72. doi: 10.1002/ppul.21558. Epub 2011 Nov 18. PMID 22102598
- [Result] Tai CC, Lu FL, Chen PC, Jeng SF, Chou HC, Chen CY, Tsao PN, Hsieh WS. Noninvasive capnometry for end-tidal carbon dioxide monitoring via nasal cannula in nonintubated neonates. Pediatr Neonatol. 2010 Dec;51(6):330-5. doi: 10.1016/S1875-9572(10)60064-2. PMID 21146797
- [Result] McSwain SD, Hamel DS, Smith PB, Gentile MA, Srinivasan S, Meliones JN, Cheifetz IM. End-tidal and arterial carbon dioxide measurements correlate across all levels of physiologic dead space. Respir Care. 2010 Mar;55(3):288-93. PMID 20196877
- [Result] Lopez E, Grabar S, Barbier A, Krauss B, Jarreau PH, Moriette G. Detection of carbon dioxide thresholds using low-flow sidestream capnography in ventilated preterm infants. Intensive Care Med. 2009 Nov;35(11):1942-9. doi: 10.1007/s00134-009-1647-5. PMID 19760396
- [Result] Cinar O, Acar YA, Arziman I, Kilic E, Eyi YE, Ocal R. Can mainstream end-tidal carbon dioxide measurement accurately predict the arterial carbon dioxide level of patients with acute dyspnea in ED. Am J Emerg Med. 2012 Feb;30(2):358-61. doi: 10.1016/j.ajem.2010.12.014. Epub 2011 Jan 28. PMID 21277140
- [Result] Howe TA, Jaalam K, Ahmad R, Sheng CK, Nik Ab Rahman NH. The use of end-tidal capnography to monitor non-intubated patients presenting with acute exacerbation of asthma in the emergency department. J Emerg Med. 2011 Dec;41(6):581-9. doi: 10.1016/j.jemermed.2008.10.017. Epub 2009 Mar 9. PMID 19272745